CLINICAL TRIAL: NCT05664100
Title: A Phase 1b, Prospective, Randomized, Single-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety of FX-345 Administered as a Single Intratympanic Injection in Adults With Acquired Adult-Onset Sensorineural Hearing Loss
Brief Title: First in Human Safety Study of FX-345 in Adults With Sensorineural Hearing Loss
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Frequency Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FX-345-101
Record Dates: First submitted 2022-12-13; First posted 2022-12-23 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Hearing loss; Intratympanic Injection
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FX-345 Cohort 1 (Experimental): Patients in the first cohort receiving FX-345 intratympanic injection
  Interventions: Drug: FX-345
- Placebo Cohort 1 (Placebo Comparator): Patients in the first cohort receiving placebo intratympanic injection
  Interventions: Drug: Placebo
- FX-345 Cohort 2 (Experimental): Patients in the second cohort receiving FX-345 intratympanic injection
  Interventions: Drug: FX-345
- Placebo Cohort 2 (Placebo Comparator): Patients in the second cohort receiving placebo intratympanic injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FX-345 — Single intratympanic injection of FX-345
  Arms: FX-345 Cohort 1; FX-345 Cohort 2
Drug: Placebo — Single intratympanic injection of placebo
  Arms: Placebo Cohort 1; Placebo Cohort 2

SUMMARY:
This single-blind, placebo-controlled trial will be conducted to evaluate the safety of FX-345 administered as a single intratympanic injection in adults with acquired sensorineural hearing loss. The primary objectives are to assess the local safety, systemic safety, and pharmacokinetic (PK) profile to determine systemic exposure.

DETAILED DESCRIPTION:
This study will enroll two cohorts. Cohort 1 (n=9) will be enrolled first to rapidly assess safety and drug exposure. After the sponsor completes an unblinded safety review, Cohort 2 (n=27) will be enrolled to continue safety evaluation of FX-345.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-67 years (inclusive)
* Documented medical history consistent with acquired, adult onset, sensorineural hearing loss
* At the Screening, Lead-in (Visit 2) and Treatment (Day 1) Visits, a pure tone average of 40- 80 dBHL at 500Hz, 1000Hz, 2000Hz, and 4000Hz in the potential study ear to be injected
* Female participants must not be pregnant, breastfeeding, or lactating. Women of child-bearing potential must agree to use a highly effective contraceptive method and must have a negative urine pregnancy test.
* Male participants must refrain from donating sperm and agree to be either abstinent or use a barrier method of contraception

Exclusion Criteria:

* Randomization in a FX-322 (laduviglusib and sodium valproate) clinical trial
* Perforation of tympanic membrane or other tympanic membrane disorders that would interfere with the delivery and safety assessment of an intratympanic medication or reasonably be suspected to affect tympanic membrane healing after injection in study ear. This includes a current tympanostomy tube.
* Any conductive hearing loss of greater than 15 dB at a single frequency or greater than 10 dB at two or more contiguous octave frequencies in the study ear at the Screening, Lead-in (Visit 2) or Treatment (Day 1) Visits, based on the investigator's judgment.
* Active chronic middle ear disease or a history of major middle ear surgery, as an adult, in the ear to be injected.
* Within 3 months of screening visit any of the following: 1) an intratympanic injection in either ear 2) treatment with steroids 3) onset of sudden sensorineural hearing loss
* Evidence of or previous diagnosis of traumatic brain injury, Meniere's disease, or genetic hearing loss
* History of head or neck radiation, significant systemic autoimmune disease, and/or chronic, recurrent clinically significant vestibular symptoms
* Exposure to another investigational drug within 28 days prior to screening visit

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Event(s) (TEAEs) | Baseline Through Day 90
Cmax | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  Maximum (peak) observed plasma drug concentration of FX04 and FX00 in cohort 1 participants
AUClast | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  Area under the concentration-time curve of FX04 and FX00 in cohort 1 participants
CL/F | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  Apparent total body clearance of FX04 and FX00 in cohort 1 participants
Vss | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  Apparent volume of distribution at steady state of FX04 and FX00 in cohort 1 participants
t1/2 | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  Elimination half-life of FX04 and FX00 in cohort 1 participants
Tmax | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  Time to reach maximum (peak) plasma drug concentration of FX04 and FX00 in cohort 1 participants
Elimination rate constant | Data points taken pre-dose and 0.5, 1, 2, 4, 6, 24 hours post-dose
  The rate at which FX04 and FX00 is removed from the human system in cohort 1 participants

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Director — Frequency Therapeutics
Locations (3):
- United States (3):
  - Clinical Trial Site, Sarasota, Florida
  - Clinical Trial Site, Spartanburg, South Carolina
  - Clinical Trial Site, San Antonio, Texas